CLINICAL TRIAL: NCT06235957
Title: Non- or Minimally Displaced Distal Radius Fractures in Adult Patients <50 Years of Age Treated Non-operatively: Three Weeks of Cast Immobilisation Versus One Week of Brace Immobilisation a Multicenter Randomised Controlled Trial.
Brief Title: Three Weeks of Cast Immobilisation Versus One Week of Brace Immobilisation in Distal Radius Fractures
Acronym: DRPIPIII
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spaarne Gasthuis (Other)
Collaborators: Maasstad Hospital (Other); Amsterdam UMC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABR 81638 | NL81638.029.22
Record Dates: First submitted 2023-11-23; First posted 2024-02-01 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Distal Radius Fractures; Fractures, Bone
Keywords: Distal radial fractures; non-operative treatment; immobilisation period
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone | interventions — POLR1G protein, human; Braces

STUDY DESIGN:
Intervention Model Description: This study will be conducted as a single-blinded multicentre randomised clinical trial in three hospitals. In this study, three weeks of cast immobilisation is compared to one week of brace immobilisation.
Who Masked: Outcomes Assessor
Masking Description: A blinded evaluation of the trial patients functional status, radiographs and range of motion will be performed by a research assistant by use of the PRWE and qDASH scores
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Other): Three weeks of cast immobilisation
  Interventions: Other: Cast 3 weeks
- Group B (Other): One week of brace immobilisation
  Interventions: Other: Brace 1 week

INTERVENTIONS:
Other: Cast 3 weeks — patients will be treated either in a cast or a brace, patients in group A are treated by cast immobilization for 3 weeks
  Arms: Group A
Other: Brace 1 week — patients will be treated either in a cast or a brace, patients in group B are treated in a brace for 1 week
  Arms: Group B

SUMMARY:
Three weeks of cast immobilisation versus one week of brace immobilisation in non- or minimally displaced distal radius fractures in adult patients <50 years of age treated non-operatively.

DETAILED DESCRIPTION:
Background: Currently, non- or minimally displaced distal radius fractures are treated by three to five weeks of cast immobilisation. Many patients with a distal radius fracture suffer from long-term functional restrictions, which might be related to stiffness due to cast immobilisation. Current literature indicates that one week of immobilisation might be safe, however, no level one evidence is available. This trial aims to compare one week of brace immobilisation with three weeks of cast immobilisation in patients with distal radius fractures that do not need reduction.

Methods: The aim of this trial is to evaluate the non-inferiority of one week of brace immobilisation in patients with non- or minimally displaced distal radius fractures. A single blinded multicentre randomised clinical trial will be conducted in three hospitals. Adult patients, between 18-50 years old, independent for activities of daily living, with a non- or minimally displaced distal radius fracture can be included in this study. The intervention group is treated with one week of brace immobilisation, and the control group with three weeks of cast immobilisation. Primary outcome is the Patient-Related Wrist Evaluation-score at six months. Secondary outcomes are: Quick Disabilities of the Arm, Shoulder and Hand-score at six weeks and six months, PRWE at six weeks, range of motion, pain, radiological outcome, complications and cost effectiveness measured by the EuroQol 5 Dimension questionnaire, Medical Consumption Questionnaire and Productivity Cost Questionnaire.

Discussion: This study will provide evidence on the optimal period of immobilisation in non-operatively treated displaced and reduced distal radius fractures. Both treatment options are accepted treatment protocols and both treatment options have a low risk of complications. Follow-up will be according to the current treatment protocol. This study will provide level one evidence on the optimal period and way of immobilisation for non- or minimally displaced distal radius fractures in adult patients.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 years (to eliminate osteoporosis);
2. Primary non- or minimally displaced DRF;
3. Independent for activities of daily living.

Exclusion Criteria:

1. Fracture of the contralateral wrist;
2. Ipsilateral fractures, proximal of the DRF;
3. Pre-existent abnormalities or functional deficits of the fractured wrist;
4. Open fractures;
5. Polytrauma patients
6. Language disability to understand the Dutch patient information and questionnaires.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Patient Related Wrist Evaluation | 6 months
  The primary outcome measure is the PRWE (Patient Related Wrist Evaluation) score after six months. Patients rate their outcome on a 0-10 scale on pain and functional outcome, and scores will be transformed to a 0-100 score. A higher score indicates greater disability.

SECONDARY OUTCOMES:
Patient Related Wrist Evaluation | 6 weeks
  The primary outcome measure is the PRWE (Patient Related Wrist Evaluation) score after six weeks The primary outcome measure is the PRWE (Patient Related Wrist Evaluation) score after six months. Patients rate their outcome on a 0-10 scale on pain and functional outcome, and scores will be transformed to a 0-100 score. A higher score indicates greater disability.
Quick Disabilities of the Arm, Shoulder and Hand | 6 weeks, 6 months
  shortened version of the DASH Outcome Measure, using 11 items instead of 30 (scored 1-5) to measure pain and functional outcome. At least 10 of the 11 items must be completed to calculate a score. The scores will be transformed to a 0-100. A higher score indicates greater disability.
Range of motion | 6 weeks, 6 months
  Range of motion measured by goniometer
Pain/Visual analogue scale score | at emergency department (day 0-1), one week, 6 weeks, 6 months
  Pain measured by VAS score VAS-score is a widely used method for pain assessments. Patients score their pain on a scale of 1-10. A higher score indicated a higher level of pain.
Radiological outcome | 6 weeks, 6 months
  Analysis of X-rays, dorsal and volar tilt in degrees, radial height in millimetres and ulnar variance in millimetres will be calculated
Complications | 6 weeks, 6 months
  Complications secondary displacement (radial shortening >3mm, dorsal tilt >10° or intra-articular step-off >2mm), delayed/non-union, re-interventions, complex regional pain syndrome (CRPS), tendon injuries (ruptures and tendinitis), nerve injuries (carpal tunnel syndrome and lesions), and distal radial ulnar joint disability.
Cost-effectiveness | 6 weeks, 6 months
  Cost-effectiveness measured by iMCQ (Medical Consumption questionnaires) Only the applicable items are included in this study. To create baseline data patients will be asked to complete those questionnaires at the ED at the day of trauma (t = 0). Patients will also be asked to complete these questionnaires at 6 weeks and 6 months
Cost-effectiveness | 6 weeks, 6 months
  Cost-effectiveness measured by iPCQ (Productivity Cost Questionnaire) Only the applicable items are included in this study. To create baseline data patients will be asked to complete those questionnaires at the ED at the day of trauma (t = 0). Patients will also be asked to complete these questionnaires at 6 weeks and 6 months
Cost-effectiveness | 6 weeks, 6 months
  Cost-effectiveness measured by EuoQol 5D (Euroquol quality of life score) Only the applicable items are included in this study. To create baseline data patients will be asked to complete those questionnaires at the ED at the day of trauma (t = 0). Patients will also be asked to complete these questionnaires at 6 weeks and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frank W Bloemers, Prof, Study Chair — Amsterdam UMC
Locations (3):
- Netherlands (3):
  - Amsterdam Umc, Amsterdam, North Holland
  - Spaarne Gasthuis, Haarlem, North Holland
  - Maasstad Ziekenhuis, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No